CLINICAL TRIAL: NCT05361863
Title: Canine Retraction Using Different Bracket Slots' Sizes: A Randomized Clinical Trial
Brief Title: Canine Retraction Using Different Bracket Slots' Sizes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Mohammed Nahidh, Principal Investigator, University of Baghdad
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 169419
Record Dates: First submitted 2022-04-30; First posted 2022-05-05 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Treating Class II Malocclusion and Bimaxillary Proclination
Keywords: Bracket slot size, canine retarction, anchorage loss
MeSH Terms: interventions — Orthodontic Brackets

STUDY DESIGN:
Intervention Model Description: The study aimed to evaluate the effectiveness of canine retraction in terms of: rate of movement and rotation using 0.020-inch slot and dual-slot systems in comparison with the 0.022-inch slot system.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The appliance and archwires will be coded for each patient, so the investigator will be blinded about the size of brackets slot and archwires gauges. Moreover, data measurements and analysis will be carried out blindly too.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 0.022×0.028-inch slot (Control Group) (Experimental): Leveling and alignment will be performed with 0.016-inch, 0.016×0.022-inch and 0.019×0.025-inch HANT followed by a working archwire of 0.019×0.025-inch stainless steel (Hangzhou Xingchen 3B Dental Instruments and Materials Co., Hangzhou, China).
  Interventions: Device: Orthodontic brackets
- 0.020×0.028-inch slot (Active Comparator): Leveling and alignment will be carried out with 0.016-inch, 0.016×0.022-inch and 0.018×0.025-inch HANT followed by a working archwire of 0.018×0.025-inch stainless steel (Hangzhou Xingchen 3B Dental Instruments and Materials Co., Hangzhou, China).
  Interventions: Device: Orthodontic brackets
- 0.018×0.028-inch slot for the anterior teeth and 0.022×0.028-inch slot for the posterior teeth (Active Comparator): Leveling and alignment will be completed with 0.016-inch, 0.016×0.016-inch, and 0.016×0.022-inch HANT followed by a working archwire of 0.016×0.022-inch stainless steel (Hangzhou Xingchen 3B Dental Instruments and Materials Co., Hangzhou, China).
  Interventions: Device: Orthodontic brackets

INTERVENTIONS:
Device: Orthodontic brackets — Interventions involving orthodontic brackets of different slot sizes

SUMMARY:
Primary Objective Evaluating the effectiveness of canine retraction in terms of: rate of movement and rotation using 0.020-inch slot and dual-slot systems in comparison with the 0.022-inch slot system.

Secondary Objectives

* Measuring the amount of molar anchorage loss during canine retraction between the different bracket slot appliances.
* Evaluation of alignment efficiency using different bracket slot appliances.

Null Hypothesis There is insignificant difference in the effectiveness of canine retraction with different bracket slot size appliances.

• Evaluation of the bracket slot and archwire dimensions precision

DETAILED DESCRIPTION:
Study Design This will be a multi-center randomized clinical trial.

Participants Participants will be recruited from subjects attending the Department of Orthodontics in the College of Dentistry, University of Baghdad and some private clinics seeking orthodontic treatment.

Sample Size Calculation Sample size will be calculated using G-power software based upon two previous trials (Mezomo et al., 2011; Moninia et al., 2019) investigating monthly canine retraction rate between conventional-ligated and self-ligating brackets. Using the highest SD and assuming the smallest difference requiring detection in canine retraction velocity to be 0.30 mm/month with an alpha level of 0.05 and power of 80%, a total of 13 canines will be required per group. Therefore, recruiting 13 patients in each group will provide 26 canines per group and this will account for dropout.

Participant Recruitment Patients seeking orthodontic treatment who meet the inclusion criteria will be assessed by the investigator for planning the orthodontic treatment. The patients will be invited to participate in the study and will be given a participant's and/or parents' information sheet to take home with them. Patients will be asked to decide about joining the trial on the next appointment (after at least one week).

Randomization and Sequence Generation Simple randomization will be accomplished with no stratification using a random number generator. A table for the allocation of the participants in the study will be composed (which includes the study number and allocation group) and kept in a sealed envelope. All the documents used for the randomization and allocation sequence generation will be kept away from the clinical environments.

Participant Allocation Numbered, identical, opaque sealed envelopes will be used for patient allocation in the current trial. The allocation envelope will contain the treatment allocation card showing either group 1, 2 or 3.

Blinding The appliance and archwires will be coded for each patient, so the investigator will be blinded about the size of brackets slot and archwires gauges. Moreover, data measurements and analysis will be carried out blindly too.

Interventions The initial records will include taking history, clinical examination, intra-oral and extra-oral photographs, dental casts, true lateral cephalograms and panoramic radiographs.

All teeth will undergo pumice and water prophylaxis immediately before bonding with a pre-adjusted edgewise fixed appliance (Hangzhou Xingchen 3B Dental Instruments and Materials Co., Hangzhou, China) MBT prescription (Table 1) with 0.022×0.028-inch slot for the first group, 0.020×0.028-inch slot for the second group and 0.018×0.028-inch slot for the anterior teeth from canine to canine and 0.022×0.028-inch slot for the posterior teeth for the third group using etching and bonding technique and light cure Transbond XT adhesive (3M Unitek, Monrovia, USA).

A standardized six-week archwire sequence (Developed by the author) will be applied for each group and as follows:

The first group with 0.022×0.028-inch slot (Control Group) Leveling and alignment will be performed with 0.016-inch, 0.016×0.022-inch and 0.019×0.025-inch HANT followed by a working archwire of 0.019×0.025-inch stainless steel (Hangzhou Xingchen 3B Dental Instruments and Materials Co., Hangzhou, China).

The second group with 0.020×0.028-inch slot Leveling and alignment will be carried out with 0.016-inch, 0.016×0.022-inch and 0.018×0.025-inch HANT followed by a working archwire of 0.018×0.025-inch stainless steel (Hangzhou Xingchen 3B Dental Instruments and Materials Co., Hangzhou, China).

The third group with 0.018×0.028-inch slot for the anterior teeth and 0.022×0.028-inch slot for the posterior teeth Leveling and alignment will be completed with 0.016-inch, 0.016×0.016-inch, and 0.016×0.022-inch HANT followed by a working archwire of 0.016×0.022-inch stainless steel (Hangzhou Xingchen 3B Dental Instruments and Materials Co., Hangzhou, China).

Before canine retraction, bondable trans-palatal arch will be inserted; omega loops will be made flush to the mesial of the buccal tube of the first molars. The second, first molars and second premolars will be tied together with stainless steel 0.010-inch ligature wire (Hangzhou Xingchen 3B Dental Instruments and Materials Co., Hangzhou, China); in addition to that the teeth from lateral incisors to its antimere on the other side will be tied too. Canine will be tied loosely with stainless steel 0.010-inch separate ligature wire and retraction will be started 28 days after insertion of the working archwire and between 7 and 14 days after extractions using NiTi closed coil spring (Hangzhou Xingchen 3B Dental Instruments and Materials Co., Hangzhou, China) tied from the first molar tube hook to the canine bracket hook using a 0.010-inch ligature wire when required to achieve the essential amount of force (about 150g) that will be checked every visit (monthly) and activated accordingly (Abu-Shahba and Alassiry, 2019).

Patients will be instructed to keep high standard oral hygiene by brushing their teeth with fluoridated toothpaste after each meal and using mouth rise when indicated.

Data Collection The following standardized data will be recorded for the trial participants before start of orthodontic treatment: full orthodontic diagnostic clinical assessment, study models, intra- and extra-oral photographs, panoramic and lateral cephalometric radiographs.

After alignment phase: digital study models, duration of alignment, rotation of canine, canine and 1st molar distance regarding the 3rd rugae, number appliance breakages.

After 4 months of canine retraction; digital study models, rate of canine movement, rotation of canine and anchorage loss.

Canines Movement Measuring canine movement will be done by projecting the distal contact point of the canine on the median palatine suture and measuring the distance from this point to the projected position of a distinct third medial rugae point in millimeters. Measurements will be made both right and left sides with the aid of AutoCAD (Figure 1). After one month, the measurements will be repeated to check reproducibility.

The total amount of movement will be considered to be the difference between the date of starting and after four months of canine retraction. The mean monthly movement was obtained by dividing the total amount of movement by the number of months during retraction (4 months).

Canines Rotation It will be represented by the angle formed between the median palatine suture and a line passing through the mesial and distal contact points of the canines Ziegler and Ingervall (1989) as shown in Figure 1.

Total rotation will be considered to be the difference between the date of starting and after four months of canine retraction. The rotation measurements will be taken after completion the alignment stage and after four months of canine retraction using AutoCAD and will be repeated after one month to check reproducibility.

Anchorage Loss The anteroposterior molar positional change will be evaluated according to the method described by Ziegler and Ingervall (1989). This will be done by projecting the mesial contact point of the first molar on the median line and measuring the distance from this point to the projected position of a distinct third medial rugae point.

Anchorage loss represented the value of subtracting the distance after four months of canine retraction from the same distance after alignment stage and for both sides. These values will be then compared among the groups. Again, measurements will be repeated using AutoCAD after one month.

Data Management A data collection sheet designed specifically for the current trial will be used to collect data from all participants' records including study models, radiographs and photographs. The data will then be analyzed by SPSS (Statistical Package for Social Sciences, IBM, NY, USA) version 25 for statistical analyses.

The following statistical tests will be used:

1. Testing the normality of data distribution by Shapiro-Wilk test.
2. Testing inter- and intra-examiner reliability by intra-class correlation coefficient test.
3. Descriptive statistics will include means, standard deviations, minimum and maximum values.
4. Inferential statistics will be represented by one-way ANOVA test followed by post hoc Tukey's test (to investigate the main study outcomes).

Withdrawal procedures Parent(s)/legal guardian(s) will be informed that they have the right to withdraw from the study at any time. The right to refuse to participate without reasons will be respected.

After the participant has entered the study, the investigator will remain free to provide alternative treatment to that specified in the protocol at any stage if he will feel that it is in the participant's best interest, but the reasons for doing so will be recorded. In these cases, the participants remain within the study for the purposes of follow-up and data analysis.

Confidentiality All participants' records will be identified in a manner designed to maintain participant confidentiality. All records will be kept in a secure storage area with limited access.

Clinical information will not be released without the written permission of the participant. Published results will not contain any personal data that could allow the identification of participants.

Dissemination of results and publication policy On completion of the trial, the data will be analyzed and a clinical study report will be prepared. In addition, the results of the trial will be presented at orthodontic national conferences and meetings. All patients recruited in the trial will be given a summary of the findings after the final report is finalized.

ELIGIBILITY:
Inclusion Criteria:

* Age 15 years and above at the start of treatment
* Molar relationship class II or I bimaxillary proclination
* Extraction of maxillary first premolar teeth as part of the orthodontic treatment
* Full set of permanent teeth regardless third molars
* No systemic diseases
* Good oral health at the start of treatment.

Exclusion Criteria:

* Orofacial clefting
* Impacted teeth
* Special needs patients
* Patients undergoing orthognathic (jaw) surgery as part of their orthodontic treatment plan
* Patients with systemic diseases requiring long-term use of Phenytoin, Cyclosporine, anti-inflammatory drugs, Bisphosphonates and systemic corticosteroids
* Poor oral hygiene, or active periodontal disease.

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
The rate of movement and/or rotation | 10 months
  Evaluating the effectiveness of canine retraction in terms of: rate of movement and/or rotation using 0.020-inch slot and dual-slot systems in comparison with the 0.022-inch slot system.

SECONDARY OUTCOMES:
Molar anchorage loss assessment during canine retraction | 10 months
  The amount of molar anchorage loss will be assessed during canine retraction among the different bracket slot appliances

CONTACTS AND LOCATIONS:
Locations (1):
- College of Dentistry, University of Baghdad, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: Undecided